CLINICAL TRIAL: NCT06672991
Title: Endoscopic Retrograde Cholangiopancreatography and Laparoscopic Cholecystectomy for Cholecystocholedocholithiasis in Children: Should It Be Accomplished in One or Repeated Hospitalization?
Brief Title: ERCP and LC for Cholecystocholedocholithiasis in Children: Should It Be Accomplished in One or Repeated Hospitalization?
Status: Completed | Type: Observational
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/30.10.2024
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Choledocholithiasis; Cholecystolithiasis; Cholangiopancreatography, Endoscopic Retrograde; Laparoscopic Cholecystectomy in Children; Children; Common Bile Duct Calculi
Keywords: Children; Endoscopic retrograde cholangiopancreatography (ERCP); Сholedocholelysis; Common Bile Duct Calculi
MeSH Terms: conditions — Choledocholithiasis; Cholecystolithiasis; Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ERCP, EST and LC in one hospitalization
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography;laparoscopic cholecystectomy
- ERCP, EST and LC on rehospitalization
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography;laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography;laparoscopic cholecystectomy — Initially, ERCP with EST was performed by an endoscopist with the consent of the patient or legal representative. The patients underwent endoscopic procedures using fluoroscopy in the operating room, under general anesthesia. Subsequently, laparoscopic cholecystectomy was performed on a delayed basis, 7 to 15 days after ERCP in a single hospitalization
  Groups: ERCP, EST and LC in one hospitalization
Procedure: Endoscopic retrograde cholangiopancreatography;laparoscopic cholecystectomy — Initially, ERCP with EST was performed by an endoscopist with the consent of the patient or legal representative. The patient underwent the endoscopic procedure using fluoroscopy in the operating room, under general anesthesia. Subsequently, laparoscopic cholecystectomy was performed on a delayed basis for readmission, 1 month after ERCP under general anesthesia.
  Groups: ERCP, EST and LC on rehospitalization

SUMMARY:
Chronic calculous cholecystitis in pediatric patients leads to choledocholithiasis in about 12% of cases. These patients require removal of stones from the common bile duct. The most common method of cleaning the common bile duct is endoscopic retrograde cholangiopancreatography, and the standard technique for removing the gallbladder is laparoscopic cholecystectomy. There are different approaches to the treatment of this category of patients: laparoscopic common bile duct exploration (LCBDE), laparoendoscopic rendezvous method (LERV) and one-stage LC after ERCP. Given the inflammation of the gallbladder and the inflammatory process in the hepatoduodenal ligament, early laparoscopic cholecystectomy can lead to various intraoperative complications. The aim of this retrospective study is to evaluate the efficacy and safety of endoscopic retrograde cholangiopancreatography, endoscopic sphincterotomy with laparoscopic cholecystectomy in a delayed manner (single or repeated hospitalization).

DETAILED DESCRIPTION:
There is no gold standard for the treatment of cholecystocholedocholithiasis in the pediatric population. The most common method for resolving biliary obstruction is endoscopic retrograde cholangiopancreatography (ERCP) with endoscopic sphincterotomy (EST) and laparoscopic cholecystectomy (LC). There are different approaches to the treatment of cholecystocholedocholithiasis: laparoscopic common bile duct exploration (LCBDE), laparoendoscopic rendezvous method (LERV) and LC after ERCP. Both LCBDE and LERV allow for the simultaneous treatment of cholecystocholedocholithiasis. However, many medical institutions do not have the opportunity to use these methods due to the difficulties of implementation and the need for specialized training and experience of specialists. The timing of LC after ERCP in patients with cholecystocholedocholithiasis remains a subject of debate. The present study aims to compare ERCP with ES + delayed LC in intra- and re-hospitalization in pediatric patients with cholecystocholedocholithiasis.

The aim of this study is to evaluate the efficacy and safety of endoscopic retrograde cholangiopancreatography, endoscopic sphincterotomy with laparoscopic cholecystectomy in a delayed manner (single or repeated hospitalization).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from child or legal guardian
* Age 0-18 years
* Acute cholecystitis
* Choledocholithiasis

Exclusion Criteria:

* Unwillingness or inability to consent to the study
* Previous ERCP or percutaneous transhepatic biliary drainage
* Benign or malignant stricture
* Preoperative comorbidities: gastrointestinal bleeding, severe liver disease, acute and chronic cholangitis, septic shock.
* In combination with Mirizzi syndrome and intrahepatic bile duct stones
* Congenital anomaly of the biliary tract
* Malignant neoplasms
* Acute pancreatitis before the procedure

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children under 18 years of age diagnosed with cholecystocholedocholithiasis
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Recurrence of common bile duct stones | 60 days after ERCP
  The diagnosis of the stone in the common bile duct was made by MRI, CT scan and ultrasound, if confirmed, before performing laparoscopic cholecystectomy.

SECONDARY OUTCOMES:
Bleeding | 30 days after ERCP
Perforation | 30 days after ERCP
  by CT, radiography (fluid or gas in the retroperitoneal space or abdominal cavity, visual picture during endoscopic examination)
Bile leak | 30 days after ERCP
  bile aspirated from the abdominal cavity
Acute cholangitis | 60 days after ERCP
  intermittent chills, fever, increased proinflammatory blood markers after ERCP
Bile duct stricture | 1 year after ERCP
  after ERCP
Time spent in hospital until discharge | from admission to hospital until the end of treatment (up to 8 weeks)
Technical success | 1 month
  - success of the procedures as documented by a yes or no
Acute pancreatitis | 30 days after ERCP
  at least two out of three criteria according to the classification developed by the INSPPIRE group
Duration of the laparoscopic cholecystectomy,min | From enrollment to the end of treatment (3 month)
Duration of the Endoscopic retrograde cholangiopancreatography,min | From enrollment to the end of treatment (3 month)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy А Pyhteev, PhD, Study Director — Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky; Leonid M Elin, Principal Investigator — Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky
Locations (1):
- Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
A complete dataset can be provided upon reasoned request